CLINICAL TRIAL: NCT03022305
Title: The Effects of Pelvic Alignment on Shoulder Range of Motion and Torque Production
Brief Title: Pelvic Alignment and Shoulder Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 201561
Record Dates: First submitted 2016-11-22; First posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Hip Alignment and Shoulder Rotation
Keywords: Hip alignment; Hip misalignment; Shoulder function; Shoulder rotation; Athletic shoulder injuries; Athletic hip alignment; Hip and shoulder alignment; Hip joint; Hip joint alignment; Hip joint misalignment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group one - standard therapy (Experimental): Standard physical therapy treatment for shoulder and hip malalignment will be administered for one week.
  Interventions: Behavioral: Group one - standard therapy
- Group two - neuromuscular therapy (Experimental): Experimental neuromuscular physical therapy treatment for shoulder and hip malalignment will be administered for one week. This therapy is exercised based.
  Interventions: Behavioral: Group two - neuromuscular therapy
- Group three - no treatment (No Intervention): No physical therapy treatment will be given to this group.

INTERVENTIONS:
Behavioral: Group one - standard therapy — Group two - standard physical therapy treatment for shoulder and hip maladjustment.
  Arms: Group one - standard therapy
Behavioral: Group two - neuromuscular therapy — Use of physical therapy treatment for shoulder and hip maladjustment.
  Arms: Group two - neuromuscular therapy

SUMMARY:
The investigators hypothesize that neuromuscular realignment of the pelvis bones will be more effective in improving range of motion and torque production at the shoulder joint than traditional exercises for improving hip internal rotation and adduction range of motion.

DETAILED DESCRIPTION:
Current literature shows a relationship between hip joint flexibility and shoulder range of motion and torque production in athletes and the general population. It is well established that limited hip joint internal rotation and adduction, specifically in baseball players, results in limited trunk rotation during pitching phase of throwing. Due to restricted rotation range at the hip joint, athletes try to compensate for the diminished rotational momentum of the trunk by producing excessive external rotation at the shoulder joint during the cocking phase of throwing. Such compensation results in laxity and overstressed shoulder joint structures. In the long term, increased laxity of the joint affects normal muscle mechanics and results in decreased torque production at the shoulder joint.

The investigators hypothesize that neuromuscular realignment of the pelvis bones will be more effective in improving range of motion and torque production at the shoulder joint than traditional exercises for improving hip internal rotation and adduction range of motion.

Group assignment:

An equal number of male and female subjects will be randomly assigned into one of three groups:

Group one will have standard treatment for improving hip range of motion. Group two will receive the new neuromuscular approach for improving pelvic alignment.

Group three will receive no treatment.

Participants and the examiners will be blinded to subjects' group assignment. Researchers will inform the subjects that they will be randomly assigned to a group with an exercise program in one of two timeframes: immediately after the initial assessment or after a one-week waiting period. Subjects in the control group will wait for one week, and then they will be asked to be tested one more time to make sure that the subject's physical condition did not change. At this time, these subjects will be informed of participation in the control group and will be given the option of going through the treatment program of choice. The neuromuscular treatment will also be offered to subjects in the standard group at the conclusion of the data collection period.

Testing procedures:

In a pretest session, the examiner, using a standard goniometer, will measure each participant's hip flexion, extension, adduction, abduction, internal rotation, and external rotation passive range of motion in seated position. Then the examiner will assess each participant's pelvic alignment using the Ober test and Thomas test. Shoulder range of motion will also be assessed using the standard goniometry procedures in the seated position. Shoulder torque production will be assessed using a Biodex isokinetic dynamometer.

The following parameters will be assessed using standard physical therapy techniques:

Hip Joint Assessment Hip range of motion assessment Hip Flexion Hip Extension Hip abduction Hip adduction Hip internal rotation Hip external rotation Ober test: [While the lower extremity is still neutral in the transverse plane, the examiner will allow the leg to slowly be lowered into full adduction. The test is considered positive if the knee joint does not reach the examination table. This test will be conducted for both sides.] Thomas test: [While holding the flexed knee to the chest, the participant will slowly lie back into a supine position on the examination table with the opposite leg hanging freely over the edge of the table. The test is considered positive if the free hanging leg is raised off the table with subject lying in supine position. This test will be conducted for both lower extremities.] Shoulder Joint Assessment Shoulder range of motion assessment Shoulder Flexion Shoulder Extension Shoulder Abduction Shoulder Internal Rotation Shoulder External Rotation Assessment of shoulder torque production: [Assessed by a Biodex isokinetic dynamometer.]

Treatment procedures:

Treatment procedure for group one:

Subjects in the standard treatment group will perform 10 repetitions of active hip internal rotation, external rotation, abduction, adduction, flexion and extension exercises daily, under supervision of the treating therapist.

Treatment neuromuscular training for group two:

Subjects in this group will perform the neuromuscular treatment for pelvic alignment, as suggested by Postural Restoration Institute, once a day under treating therapist supervision for one week. Subject will flex the hip and knee joints to 90° and will rest both feet against the wall with a standard 4 - 6" ball will be placed between the subject's knees. At this position, the subject is instructed to squeeze the ball between the knees and to perform an isometric hamstring muscle contraction (statically pulling the feet downward without pressing to the wall). At this point, the subject will be instructed to perform a gentle posterior pelvic tilt while avoiding abdominal muscle contraction. While maintaining this position, the subject is instructed to take a deep breath in through the nose and then slowly blow out into the balloon. The subject will be instructed to pause for 3 seconds while pressing the tongue to the roof the mouth to prevent airflow out of the balloon. After the 4th breath in, the subject will pinch the neck of the balloon and remove it from the mouth. Then subject will relax and take the feet off the wall. This exercise will be repeated daily for one week (Monday through Friday). Following neuromuscular training exercise, the patient will perform a coordinated hip internal and external rotation exercise in side lying.

The no treatment group will act as a control group. Both the standard and no treatment group will be offered free neuromuscular treatment at the conclusion of posttest data collection.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria includes:

  * College-aged students between the ages of 18 and 25,
  * Having limited hip ROM than the normal ranges suggested by the AAOS guidelines,
  * Having positive Ober and Thomas tests,

Exclusion Criteria:

* Exclusion criteria is as follows:

  * Having known shoulder pathologies,
  * Structural leg length discrepancies,
  * Having any cardiovascular, respiratory or other health problems
  * Require use of an assistive device for ambulation,
  * Amputees, and people with structural deformities of the shoulder or hip joint.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pelvic realignment achieved as indicated by negative Ober test on examination at completion of the training period.. | Outcomes will be assessed following one week for each of the therapy groups.
  Results of the three groups, (1) standard conditioning, (2) neuromuscular conditioning, and (3) no conditioning, will be assessed for pelvic realignment following one week of each of these therapies.

SECONDARY OUTCOMES:
Pelvic realignment achieved as indicated by negative Thomas test on examination at completion of the training period.. | Outcomes will be assessed following one week for each of the therapy groups.
  Results of the three groups, (1) standard conditioning, (2) neuromuscular conditioning, and (3) no conditioning, will be assessed for pelvic realignment following one week of each of these therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Nourbakhsh, PhD, Principal Investigator — University of North Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robb AJ, Fleisig G, Wilk K, Macrina L, Bolt B, Pajaczkowski J. Passive ranges of motion of the hips and their relationship with pitching biomechanics and ball velocity in professional baseball pitchers. Am J Sports Med. 2010 Dec;38(12):2487-93. doi: 10.1177/0363546510375535. Epub 2010 Aug 31. PMID 20807860
- [Background] Edouard P, Samozino P, Julia M, Gleizes Cervera S, Vanbiervliet W, Calmels P, Gremeaux V. Reliability of isokinetic assessment of shoulder-rotator strength: a systematic review of the effect of position. J Sport Rehabil. 2011 Aug;20(3):367-83. doi: 10.1123/jsr.20.3.367. PMID 21828388
- [Background] Baltaci G, Tunay VB. Isokinetic performance at diagonal pattern and shoulder mobility in elite overhead athletes. Scand J Med Sci Sports. 2004 Aug;14(4):231-8. doi: 10.1111/j.1600-0838.2004.00348.x. PMID 15265145
- [Result] Laudner K, Wong R, Onuki T, Lynall R, Meister K. The relationship between clinically measured hip rotational motion and shoulder biomechanics during the pitching motion. J Sci Med Sport. 2015 Sep;18(5):581-4. doi: 10.1016/j.jsams.2014.07.011. Epub 2014 Jul 30. PMID 25130280